CLINICAL TRIAL: NCT05912543
Title: A Titration of Fractional Inspired Oxygen Using Oxygen Reserve Index (ORi™) During One-lung Ventilation in the Pediatric Patient: a Randomized Controlled Trial
Brief Title: A Titration of Fractional Inspired Oxygen Using Oxygen Reserve Index in Child
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ji-Hyun Lee, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2205-156-1329
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2023-06

CONDITIONS: Hyperoxemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional arm (No Intervention): Moderate hyperoxia as determined by T1 arterial blood gas. For moderate hyperoxemia (PaO2 > 300 mmHg), reduce the inspired oxygen concentration to 80% and for severe hyperoxemia to 70%.
  In the situation of hypoxia, where the peripheral oxygen saturation decreases to less than 95% even in 100% of FiO2, the following treatment is indicated: Fluid administration, inotropes administration (dopamine), alveolar recruitment, return to two-lung ventilation, and application of continuous positive airway pressure.
- ORI arm (Experimental): Target ORi™ of 0.15, check the ORi™ every 5 minutes and adjust the inspired oxygen concentration in 5% increments. If the ORi™ decreases to less than 0.15, treat it in the same way as if hypoxia occurred in the conventional group.
  Interventions: Procedure: Titration of FiO2

INTERVENTIONS:
Procedure: Titration of FiO2 — The inhaled oxygen concentration after one-lung ventilation will be treated by the group.
  Arms: ORI arm

SUMMARY:
The purpose of this prospective randomized controlled trial is to determine whether using the Oxygen Reserve Index can prevent hyperoxemia in pediatric patients receiving single-lung ventilation.

Participants will have their FiO2 adjusted in a prescribed manner based on the arm to which they are assigned.

The researchers will compare whether blood oxygen levels were lower in the ORI group.

ELIGIBILITY:
Inclusion Criteria:

* Children under 7 years of age undergoing surgery under unilateral pulmonary ventilation
* Children with American Society of Anesthesiology physical status I, II, III

Exclusion Criteria:

* Patient who have chronic respiratory failure
* Patient who have a history of bronchopulmonary dysplasia, respiratory distress syndrome of neonate, laryngomalacia, tracheomalacia or tracheal stenosis
* Patient whose initial Oxygen Reserve Index value is zero
* Patient who need supplementary oxygen before surgery

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2023-06-25 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
The incidence of moderate to severe hyperoxemia in arterial blood gas analysis at T2 (30 minutes after one lung ventilation) | 30 minutes after initiation of one-lung ventilation
  arterial oxygen content over 200

SECONDARY OUTCOMES:
average Oxygen Reserve Index value | during one lung ventilation
time-weighted average inspired oxygen fraction | during one lung ventilation
incidence of hypoxemia | perioperative period
incidence of perioperative complications | perioperative period

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No